CLINICAL TRIAL: NCT04014218
Title: Effect of Inhalation Sedation With Sevoflurane Compared With Propofol on the Sepsis-related Acute Respiratory Distress Syndrome (ARDS) Course.
Brief Title: Effect of Inhalation Sedation Compared With Propofol on the Sepsis-related Acute Respiratory Distress Syndrome Course
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Valery V. Likhvantsev, Professor, Professor, Head of Intensive Care Department Moscow Regional Clinical and Research Institute, Moscow Regional Research and Clinical Institute (MONIKI)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SS2019
Record Dates: First submitted 2019-07-02; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: ARDS
Keywords: sedation; ARDS; sepsis; outcome
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: opaque envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhalation sedation (Experimental)
  Interventions: Drug: Inhalation Sedation
- Propofol (Active Comparator)
  Interventions: Drug: Intravenous Sedation

INTERVENTIONS:
Drug: Inhalation Sedation — Inhalation Sedation by Administration of Sevoflurane
  Arms: Inhalation sedation
Drug: Intravenous Sedation — Intravenous Sedation by Administration of Propofol
  Arms: Propofol

SUMMARY:
Investigation of effect of inhalation sedation by administration of Sevoflurane compared with Propofol on the moderate acute respiratory distress syndrome course in mechanically ventilated patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* sepsis
* ARDS
* P/F Ratio 100-250
* start of mechanical ventilation

Exclusion Criteria:

* pregnancy
* concomitant oncological disease
* prior psychological impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 days after ICU admission
  28 days and in-hospital mortality
ICU Length of stay (LOS) | 45 days after ICU admission
  Length of stay in ICU
Length of mechanical ventilation (LMV) | 45 days after ICU admission
  Length of mechanical ventilation

SECONDARY OUTCOMES:
P/F Ratio | 45 days after ICU admission
  minimal pO2/FiO2
Delirium | 5 days after ICU admission
  onset and duration of delirium
MACCE | 28 days after ICU admission
  Major Adverse Cardiac and Cerebrovascular Event
event of RRT | 28 days after ICU admission
  event of Renal Replacement Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Valery V Likhvantsev,, Principal Investigator — Moscow Regional Clinical and Research Institute, Department of Intensive Care
Locations (1):
- Moscow Regional Research and Clinical Institute Moniki n.a. M.F. Vladimirskiy, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No